CLINICAL TRIAL: NCT00986583
Title: Effect of Succinylcholine on Patients Using Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Alparslan Turan, Principal Investigator, The Cleveland Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-683
Record Dates: First submitted 2009-09-23; First posted 2009-09-30 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Pain
Keywords: Succinylcholine; Statins; myalgias; statins with succinylcholine and pain
MeSH Terms: conditions — Pain; Myalgia | interventions — Succinylcholine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Statin use group (Other): Patients taking simvastatin, lovastatin, atorvastatin, or pravastatin for at least three months.
  Interventions: Drug: Succinylcholine
- non statin use (Other): Patients not taking simvastatin, lovastatin, atorvastatin, or pravastatin for at least three months.
  Interventions: Drug: Succinylcholine

INTERVENTIONS:
Drug: Succinylcholine — Succinylcholine will be administered pre-induction over a period of 5 seconds

SUMMARY:
Based on available mechanistic and clinical information, the investigators propose a nonrandomized study to evaluate the effect of succinylcholine in patients taking statins. The investigators' purpose is to evaluate the effect of succinylcholine on patients taking statins. Patients scheduled to undergo elective surgery (other then orthopedic, spinal, vascular or muscle) with planned endotracheal intubation will be approached regarding participation in the trial. Design of the study is complex because there is no way to randomize patients to statins or no statins and also no way to take them off the statins prior surgery. So statin use will not be randomized; confounding factors will be accounted for by stratification (every 10 years of age from 40-80 and gender) and statistical adjustment. The investigators propose to test the hypothesis that succinylcholine administration increases plasma myoglobin concentration more in patients who are on statins compared to patients who do not.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery not involving orthopedic procedure, muscle and spinal surgery
* ASA Physical Status 1-3

Exclusion Criteria:

* History of liver failure
* History of renal failure
* History of neuromuscular disease
* Increased intraocular pressure
* Recent major burn
* Multiple trauma
* Susceptibility to or family history of malignant hyperthermia

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alparsan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients taking simvastatin, lovastatin, atorvastatin, or pravastatin for at least 3 months and those who had never used statins were considered to be eligible for participation. We included patients scheduled for elective surgery (October 2009 between June 2010) in this comparative, prospective, nonrandomized study.
Period: Overall Study
Arm/Group | Statin Use Group | Non Statin Use
Started | 38 | 32
Completed | 38 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Statin Use Group | Non Statin Use | Total
Number analyzed (Participants) | 38 | 32 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9) | 57 (10) | 59 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 22 | 17 | 39
Region of Enrollment [Number; unit: participants]
  United States | 38 | 32 | 70

OUTCOME MEASURES:

1. Primary Outcome: Plasma Myoglobin Concentration
Time Frame: induction, 5 minutes after administration, 20 minutes and 24 hours post operatively
Measure: Median (Inter-Quartile Range); unit: ug/l
Arm/Group | Statin Use Group | Non Statin Use
Number analyzed (Participants) | 38 | 32
ug/l
  Measurement time = induction (0 minute) | 46 [40 to 59] | 39 [29 to 49]
  Measurement time = 5 minute | 71 [47 to 96] | 49 [31 to 75]
  Measurement time = 20 minute (primary) | 77 [49 to 112] | 47 [35 to 79]
  Measurement time = 24 hour | 137 [86 to 342] | 95 [57 to 210]
Statistical Analysis 1: Comparison: Statin Use Group vs Non Statin Use; Test type: Superiority or Other; p = 0.018, ANCOVA — This is for the primary comparison at 20 minute; Ratio of medians = 1.34, 95% CI 2-sided [1.05 to 1.72] — Ratio of medians of myoglobin measured at 20 minute for statin users vs. non-statin users

2. Secondary Outcome: Muscle Pain
Description: verbal rating scale score and the pain score both at 2 and 24 hours postoperatively.
  The verbal rating scale score ranges from 0 (no pain) to 100 (worst pain imaginable).
  The pain score ranges from 0 to 3: 0 none; 1 muscle stiffness or pain in the nape of the neck, shoulders, and chest; 2 muscle stiffness and pain requiring analgesia; and 3 incapacitating generalized muscle stiffness or pain.
Time Frame: 2 and 24 hours postoperatively
Measure: Number; unit: participants
Arm/Group | Statin Use Group | Non Statin Use
Number analyzed (Participants) | 38 | 32
participants
  VRS score at 2 hour: 0 (no pain) | 34 | 26
  VRS score at 2 hour: 10-30 | 2 | 0
  VRS score at 2 hour: 40-70 | 1 | 4
  VRS score at 2 hour: 80-100 | 1 | 2
  VRS score at 24 hour: 0 (no pain) | 34 | 25
  VRS score at 24 hour: 10-30 | 2 | 4
  VRS score at 24 hour: 40-70 | 1 | 2
  VRS score at 24 hour: 80-100 | 1 | 1
  Pain score at 2 hour: 0 (no pain) | 34 | 26
  Pain score at 2 hour: 1 | 4 | 3
  Pain score at 2 hour: 2 | 0 | 3
  Pain score at 24 hour: 0 (no pain) | 34 | 25
  Pain score at 24 hour: 1 | 4 | 5
  Pain score at 24 hour: 2 | 0 | 2

3. Secondary Outcome: Serum Potassium Concentration
Time Frame: At 5 and 20 min after succinylcholine
Population: Two patients in non-statin group had missing value at 20 minute.
Measure: Median (Inter-Quartile Range); unit: mEq/l
Arm/Group | Statin Use Group | Non Statin Use
Number analyzed (Participants) | 38 | 30
mEq/l
  at 5 minute | 4.2 [4.0 to 4.5] | 4.2 [4.0 to 4.5]
  at 20 minute | 4.0 [3.7 to 4.3] | 3.9 [3.7 to 4.1]

4. Secondary Outcome: Change in Plasma Creatine Phosphokinase (CK) Concentration From 2 to 24 Hours Postoperatively
Description: Change in plasma creatine phosphokinase (CK) concentration from 2 to 24 hours postoperatively
Time Frame: 2 and 24 hours postoperatively
Population: Two patients in the nonstatin group had missing CK value at 2 hour
Measure: Median (Inter-Quartile Range); unit: units/l
Arm/Group | Statin Use Group | Non Statin Use
Number analyzed (Participants) | 38 | 30
units/l | 175 [11 to 333] | 78 [19 to 354]

5. Secondary Outcome: Duration of Succinylcholine Block
Description: Time required to reach maximum block by succinylcholine after succinylcholine administration.
Time Frame: intraoperative: from succinylcholine administration
Measure: Median (Inter-Quartile Range); unit: minute
Arm/Group | Statin Use Group | Non Statin Use
Number analyzed (Participants) | 38 | 32
minute | 4.2 [3.0 to 6.0] | 4.6 [3.3 to 6.1]

6. Secondary Outcome: Fasciculation
Description: The fasciculation ranges from 0 to 3: 0 none; 1 small movements around eyes and fingers; 2 moderate movements in face, neck, fingers, and trunk; and 3 vigorous movements in trunk and extremities.
Time Frame: postoperative
Measure: Number; unit: participants
Arm/Group | Statin Use Group | Non Statin Use
Number analyzed (Participants) | 38 | 32
participants
  None | 9 | 13
  Small | 6 | 3
  Moderate | 10 | 8
  Vigorous | 13 | 8

ADVERSE EVENTS:
Arm/Group | Statin Users | Nonstatin Users
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/32
Other Adverse Events (participants affected / at risk) | 0/38 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes